CLINICAL TRIAL: NCT06223932
Title: Evaluation of the Efficacy and Safety of Molnupiravir Treatment in Mild/Moderate Covid-19 Patients. Turkey Cohort, Prospective, Observational, Comparative Study
Brief Title: Evaluation of the Efficacy and Safety of Molnupiravir Treatment in Mild/Moderate Covid-19 Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Serap Yavuz (Other)
Collaborators: MDX Klinik Araştırma Egitim ve Danismanlik Ltd. Sti. (Unknown)
Responsible Party: Sponsor-Investigator, Serap Yavuz, Prof. MD., Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: 11881
Record Dates: First submitted 2024-01-23; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Infection; Molnupiravir; 11881; Istanbul University, Department of Infectious Disease
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 diagnosed patients receiving molnupiravir: COVID-19 diagnosed patients receiving molnupiravir treatment
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Molnupiravir — COVID-19 diagnosed patients receiving molnupiravir will be evaluated to show if Molnupiravir is effective in reducing the combined outcome of hospitalization/death due to COVID-19 in the first 28 days when used in real life.

SUMMARY:
Evaluation of the Efficacy and Safety of Molnupiravir Treatment in Mild/Moderate Covid-19 Patients. Turkey Cohort, Prospective, Observational, Comparative Study In the antiviral treatment of COVID-19, molnupiravir, an RdRp (RNA-dependent RNA polymerase) inhibitor, was the first agent shown to reduce death and hospitalization in a reliable/adequate phase-3 clinical trial. For this reason, molnupiravir has been approved for emergency use in many countries, including Turkey, as it is still an unmet need in the treatment of COVID-19. However, it is not yet known which factors related to the patient or the disease are important for this drug to be effective. In addition, since this is the first time it will be widely used, rare or long-term adverse effects have not been identified. Since molnupiravirin is known to exert antiviral activity by inducing mutations in the virus, there are some hypotheses that this effect may lead to the emergence of new and more dangerous variants.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether molnupiravir, which will be used as the first antiviral drug outside of the repositioned options in the treatment of COVID-19, is effective in reducing the combined outcome of hospitalization/death due to COVID-19 in the first 28 days when used in real life. (Note: In patients diagnosed with COVID-19 while hospitalized for other reasons and included in the study, COVID-19-related oxygen requirement + COVID-19-related death will be considered as the primary outcome).

The secondary objectives of this study are as follows:

1. Molnupiravirin in COVID-19 patients,

   1. Clinical improvement on days 3, 5, 10, 14 and 28 (according to the WHO clinical status assessment scale)
   2. On oxygen requirement in the first 28 days,
   3. On the need for ICU in the first 28 days,
   4. On the need for ventilatory support in the first 28 days,
   5. Viral clearance rates on days 3, 5, 10 and 14,
   6. On day 10, on serum glucose, BUN, creatinine, AST, ALT, CRP, LDH, procalcitonin, D-Dimer levels, blood leukocyte, neutrophil and lymphocyte, erythrocyte and platelet counts
   7. On mortality rates at 28 days and 3 months
   8. Adverse drug effects seen at 3rd, 5th, 10th, 14th days, 28 days, 3rd and 6th months, analysis of the effects
   9. Monitoring the patient's general condition and new disease diagnoses at 3 and 6 months
2. In COVID-19 patients receiving molnupiravir, 10) Identification of the presence and proportion of mutant SARS-CoV-2 present in day 5, 10 and 14 samples 11) Determination of the ratio of those who grow in viral culture and those who may be infectious in people whose SARS-CoV-2 positivity was detected in samples on the 5th, 10th and 14th days 12) Determination of the phenotypic susceptibility of SARS-CoV-2 strains to molnupiravir in samples collected on days 5, 10 and 14
3. Determining which factors are associated with the efficacy of molnupiravir in reducing hospitalization and mortalitySince it is known that molnupiravir has antiviral activity by inducing mutation in the virus, there are some hypotheses that this effect may lead to the emergence of new and more dangerous variants.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity (BMI >30 kg/m2 in adults), chronic renal failure, diabetes mellitus, presence of immunosuppressive diseases or drug use, cardiovascular diseases (including congenital heart diseases or hypertension), chronic lung diseases, among the comorbidities that cause severe Covid-19; (e.g. COPD, moderate to severe asthma, cystic fibrosis, interstitial lung disease, pulmonary hypertension, chronic liver disease concomitant to nonconcomitant cirrhosis), neurological developmental diseases (e.g. cerebral palsy), sickle cell anemia, other medical complex conditions (e.g. genetic or metabolic syndromes or severe congenital anomalies) and
2. Positive SARS-CoV-2 PCR test or SARS-CoV-2 rapid antigen test in nasopharyngeal swab specimen,
3. Have at least 1 symptom consistent with COVID-19,
4. No more than 5 days have elapsed since the onset of symptoms,
5. Outpatients or those diagnosed with COVID-19 while hospitalized for reasons other than COVID-19,
6. Those for whom molnupiravir treatment is recommended in the current COVID-19 Treatment Guidelines of the Ministry of Health.

Exclusion Criteria:

1. <18 years old
2. Pregnant or breastfeeding
3. Patients whom the researcher thinks may have problems with compliance,
4. Patients with an increased need for oxygen due to COVID-19
5. Patients receiving corticosteroid or anti-cytokine therapy for COVID-19,
6. Patients >5 days from the onset of symptoms
7. Subjects with chronic diarrhea or chronic gastrointestinal problems that may impair drug absorption,
8. History of allergy to molnupiravir,
9. Those with chronic alcoholism
10. Those who have received another antiviral therapy targeting SARS-CoV-2 (favipiravir, remdesivir, specific monoclonal antibodies, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 18-65 years old patients
  * Patients with a confirmed diagnosis of COVID-19 who were offered and accepted molnupiravir treatment by their attending physician: 1300 patients
  * Patients with a confirmed diagnosis of COVID-19 who were offered molnupiravir treatment by the attending physician and refused to take it: 1300 patients
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Molnupiravir effectineness in reducing the combined outcome of hospitalization/death due to COVID-19 in the first 28 days when used in real life | 28 Days, 3 month and 6 month follow-up after diagnose and treatment
  The primary objective of this study is to determine whether molnupiravir, which will be used as the first antiviral drug outside of the repositioned options in the treatment of COVID-19, is effective in reducing the combined outcome of hospitalization/death due to COVID-19 in the first 28 days when used in real life. (Note: In patients diagnosed with COVID-19 while hospitalized for other reasons and included in the study, COVID-19-related oxygen requirement + COVID-19-related death will be considered as the primary outcome).

CONTACTS AND LOCATIONS:
Locations (8):
- Turkey (Türkiye) (8):
  - Istanbul University, Istanbul Faculty of Medicine, Department of Infectious Disease, Istanbul, Fatih
  - Cerrahpasa Faculty of Medicine Infectious Disease Departament, Istanbul, Fatih
  - Ankara City Hospital, Ankara
  - Ankara University Faculty of Medicine, Ankara
  - CAM and SAKURA Training and Research Hospital, Istanbul
  - Istanbul Haseki Training and Research Hospital, Istanbul
  - Koc University Hospital, Istanbul
  - Umraniye Training and Research Hospital, Istanbul